CLINICAL TRIAL: NCT05484193
Title: Comparison of Pregnancy Rates After Luteal Phase Support With GnRH Agonist Versus Progesterone - a Prospective Randomized Study
Brief Title: GnRH Agonist for Luteal Phase Support.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Synarel fresh LPS
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Use of GnRH Agonist Alone for Luteal Phase Support in Fresh IVF Cycles
MeSH Terms: interventions — Gonadotropin-Releasing Hormone; Nafarelin; Progesterone; Utrogestan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GnRH-agonist group (Experimental): In the GnRH-a group, LPS was initiated on the evening after the OPU, using Nafareline (Synarel nasal spray 200mg used once), followed by twice daily (total 400mg/day) until the day of serum β-hCG pregnancy test, and then stopped, regardless of the test results
  Interventions: Drug: GnRH agonist
- Progesterone group (Active Comparator): In the progesterone group, LPS was initiated on the morning after OPU, using micronized progesterone ( PV Utrogestan 300mg, 3 times daily), until serum β-hCG pregnancy tests results were available. If a β-hCG pregnancy was confirmed, LPS was continued until the end of the 8th gestational week
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: GnRH agonist — GnRH agonist alone for luteal phase support in fresh IVF embryo transfer cycles
  Other Names: Synarel
  Arms: GnRH-agonist group
Drug: Progesterone — vaginal progesterone for luteal phase support
  Other Names: Utrogestan
  Arms: Progesterone group

SUMMARY:
Objective To assess the the efficacy of luteal support with GnRH agonist in patients undergoing IVF in antagonist-based hcg triggered cycles compared with standard luteal support with progesterone.

Design prospective randomized controled study Subjects Patients who underwent antagonist-based cycles performed in the "Shaare Zedek Medical Center" IVF clinic between 2020 and 2022 Intervention Intranasal GnRH-agonist or vaginal Progesterone for luteal support.

Main outcome measures Pregnancy and clinical pregnancy rates, ohss.

The study cohort included 150 patients who underwent 164 cycles. A total of 127 cycles were included. Of them, 64 were treated with GnRH-a and 63 with progesterone.

Hypothesis: This RCT suggests that GnRH-a for luteal phase support is associated with a higher positive β-hCG pregnancy rate and clinical pregnancy rate, compared with standard progesterone support in an antagonist-based protocol triggered with hCG, while maintaining a similar safety profile.

ELIGIBILITY:
Inclusion Criteria:Criteria for inclusion were patients aged between 18-45 years, BMI between 19-35, infertility diagnosis of male factor, tubal factor, anovulation, unexplained and age-related. Patients with or without infertility diagnosis, who underwent IVF for PGT were also included.

-

Exclusion Criteria:

Exclusion criteria were triggering with agents other than hCG, previous 3 or more failed cycles in which a good quality embryo or embryos were transferred, endometriosis, hydrosalpinx, hypogonadotropic hypogonadism, and Mullerian malformations. Drop-out criteria included no fresh embryo transfer, intolerance to GnRH-a, and nasal congestion during the luteal phase.

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
pregnancy | 2 weeks
  - positive Bhcg

SECONDARY OUTCOMES:
clinical pregnancy | 5 weeks
  gestational sac with heartbeat
ovarian hyperstimulation syndrome | 5 weeks
  early and late

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Buhbut E, Nabulsi R, Avigdor G, Ben-Ami I. Comparison of pregnancy rates in antagonist cycles after luteal support with GnRH-agonist versus progesterone: prospective randomized study. Arch Gynecol Obstet. 2023 Jul;308(1):255-263. doi: 10.1007/s00404-023-07017-5. Epub 2023 Apr 25. PMID 37186265